CLINICAL TRIAL: NCT01369329
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Safety and Efficacy of Ustekinumab Induction Therapy in Subjects With Moderately to Severely Active Crohn's Disease Who Have Failed or Are Intolerant to TNF Antagonist Therapy (UNITI-1)
Brief Title: A Study to Evaluate the Safety and Efficacy of Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease Who Have Failed or Are Intolerant to Tumor Necrosis Factor (TNF) Antagonist Therapy (UNITI-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018415; CNTO1275CRD3001 (Other: Janssen Research & Development, LLC); 2010-022758-18 (EudraCT Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Crohn's Disease; IBD; Colitis; Inflammatory Bowel Disease
Keywords: ustekinumab; moderately to severely active Crohn's Disease; tumor necrosis factor, Stelara; Crohn; Crohn's; IBD; UNITI
MeSH Terms: conditions — Crohn Disease; Colitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 001 (Placebo Comparator): Group 1: Placebo Form=solution for injection route=intravenous use in a single dose.
  Interventions: Drug: Group 1: Placebo
- 002 (Experimental): Group 2 ustekinumab 130 mg Type=exact unit=mg number=130 form=solution for injection route= intravenous use in a single dose.
  Interventions: Drug: Group 2 ustekinumab 130 mg
- 003 (Experimental): Group 3: ustekinumab approximately 6 mg/kg Type=range unit=mg/kg number=6 form=solution for injection route= intravenous use in a single dose.weight-range based ustekinumab doses approximating ustekinumab 6 mg/kg: 260 mg (weight <= 55 kg) 390 mg (weight > 55 kg and <= 85 kg) and 520 mg (weight > 85 kg).
  Interventions: Drug: Group 3: ustekinumab approximately 6 mg/kg

INTERVENTIONS:
Drug: Group 2 ustekinumab 130 mg — Type=exact, unit=mg, number=130, form=solution for injection, route= intravenous use, in a single dose.
  Arms: 002
Drug: Group 3: ustekinumab approximately 6 mg/kg — Type=range, unit=mg/kg, number=6, form=solution for injection, route= intravenous use, in a single dose.weight-range based ustekinumab doses approximating ustekinumab 6 mg/kg: 260 mg (weight <= 55 kg), 390 mg (weight > 55 kg and <= 85 kg), and 520 mg (weight > 85 kg).
  Arms: 003
Drug: Group 1: Placebo — Form=solution for injection, route=intravenous use, in a single dose.
  Arms: 001

SUMMARY:
This study (UNITI-1) will compare the effects (both positive and negative) of an initial treatment with ustekinumab to placebo over 8 weeks, in patients with moderately to severely active Crohn's disease who have either failed or could not tolerate at least one TNF-antagonist medications in the past (specifically, infliximab, adalimumab, or certolizumab pegol).

DETAILED DESCRIPTION:
This study (CNTO1275CRD3001 or "UNITI-1") examines ustekinumab (an antibody medication that inhibits the inflammatory proteins IL-12 and IL-23) versus a placebo (otherwise identical except without the ustekinumab antibody) given intravenously (by an IV) in adults with moderately to severely active Crohn's disease who previously did not respond to, lost response to, or could not tolerate TNF-antagonist medications (specifically, infliximab, adalimumab or certolizumab pegol). Ustekinumab (also known as Stelara) is approved as a treatment for the skin condition of moderate to severe plaque-type psoriasis, but this study will examine if ustekinumab can provide benefit in Crohn's disease and also assess for any risks or side effects. Both the positive and negative outcomes of IV placebo versus two different doses of IV ustekinumab will be tracked and compared over eight weeks, in approximately 703 patients. Patients enrolling in this study will be assigned to one of the 3 treatment groups by chance (randomly, like rolling dice), and all will receive a single IV administration of study agent at the first study visit (after the screening period), and then will be asked to return for 3 additional visits through Week 8. Patients who complete this study through the Week 8 visit and remain eligible can enter the maintenance study (CNTO1275CRD3003 or "IM-UNITI'' [NCT01369355]), where they will receive additional study agent, including the administration of ustekinumab in patients who receive placebo in this study and have not had improvement in their Crohn's disease. Patients who do not enter the CNTO1275CRD3003 study will have a final safety follow-up visit approximately 20 weeks after they received study agent when they entered into this study at the Week 0 visit. .All patients will receive a single intravenous (IV) administration of study drug (either placebo or ustekinumab) at the first (week 0) visit when they enter the study.There are 3 treatment groups: Group 1: Placebo; Group 2: ustekinumab 130 mg, Group 3: weight-range based ustekinumab doses approximating ustekinumab 6 mg/kg: 260 mg (weight <= 55 kg), 390 mg (weight > 55 kg and <= 85 kg), and 520 mg (weight > 85 kg).

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease of at least 3 months' duration with colitis, ileitis, or ileocolitis, confirmed at some time in the past by radiography, histology, or endoscopy
* Have active Crohn's disease, defined as a baseline Crohn's Disease Activity Index (CDAI) score of >= 220 and <= 450
* Have received infliximab, adalimumab, or certolizumab pegol at a dose approved for the treatment of Crohn disease and did not respond initially (ie, primary nonresponse)
* Or responded initially but then lost response with continued therapy (ie, secondary nonresponse)
* Or were intolerant to the medication
* Have screening laboratory test results within protocol-specified parameters.

Exclusion Criteria:

* Patients who have had any kind of bowel resection within 6 months
* Are pregnant or planning pregnancy (both men and women) while enrolled in the study or for 20 weeks after receiving study agent
* Patients who have received infliximab, adalimumab or certolizumab pegol < = 8 weeks before the first administration of study drug
* Patients with certain complications of Crohn's disease that would make it hard to assess response to study drug
* Patients with a history of or ongoing chronic or recurrent infectious disease
* Patients who have previously received a biologic agent targeting IL-12 or IL-23, including but not limited to ustekinumab (CNTO 1275) or briakinumab (ABT-874)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (175):
- United States (67):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - Redwood City, California
  - San Carlos, California
  - San Diego, California
  - Lone Tree, Colorado
  - New Haven, Connecticut
  - Gainesville, Florida
  - Jacksonville, Florida
  - Weston, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - Clive, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Novi, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Ocean Springs, Mississippi
  - Lees Summit, Missouri
  - Urbana, Missouri
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Marlton, New Jersey
  - Morristown, New Jersey
  - Great Neck, New York
  - New York, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Beavercreek, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Springfield, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - North Charleston, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (8):
  - Bedford Park
  - Box Hill
  - Central Queensland M C
  - Concord
  - Garran
  - Liverpool
  - Malvern
  - Parkville
- Austria (3):
  - Innsbruck
  - Sankt Pölten
  - Vienna
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Rio de Janeiro, Brazil
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brandon, Manitoba
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Montreal, Quebec
- Czechia (2):
  - Hradec Králové
  - Ústí nad Labem
- Denmark (2):
  - Herlev
  - Silkeborg
- France (10):
  - Amiens
  - Caen
  - Lille
  - Marseille
  - Nantes
  - Paris
  - Pessac
  - Reims
  - Rouen
  - Toulouse
- Germany (19):
  - Berlin
  - Erlangen
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Jena
  - Kiel
  - Lÿneburg
  - Mannheim
  - Minden
  - München
  - Münster
  - Regensburg
  - Tübingen
  - Ulm
- Szekszárd, Hungary
- Iceland (2):
  - Akureyri
  - Reykjavik
- Dublin, Ireland
- Israel (2):
  - Jerusalem
  - Tel Litwinsky
- Japan (12):
  - Chikushino-shi
  - Fukuoka
  - Hamamatsu
  - Kagoshima
  - Nishinomiya
  - Ohtsu
  - Osaka
  - Ōita
  - Sakura
  - Sapporo
  - Tokyo
  - Yokkaichi
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Rotterdam
- New Zealand (4):
  - Auckland
  - Christchurch
  - Grafton
  - Hamilton
- Poland (2):
  - Krakow
  - Lodz
- Serbia (2):
  - Belgrade
  - Niš
- South Africa (2):
  - Cape Town
  - Overport
- Seoul, South Korea
- Spain (2):
  - Madrid
  - Sagunto
- United Kingdom (17):
  - Birmingham
  - Brighton
  - Bristol
  - Cambridge
  - Cardiff
  - Exeter
  - Gloucester
  - Harrow
  - Liverpool
  - London
  - Manchester
  - Norwich
  - Nottinghamshirecc
  - Oxford
  - Shropshire
  - South Shields
  - Southampton

REFERENCES:
- [Derived] Huan PW, Mehta A, Wong ECL, Dulai PS, Marshall JK, Reinisch W, Narula N. A Review of the Modified Multiplier of Simple Endoscopic Score for Crohn's Disease and How to Use It in Clinical Trials and Practice. Am J Gastroenterol. 2025 Oct 1;120(10):2242-2250. doi: 10.14309/ajg.0000000000003373. Epub 2025 Feb 25. PMID 39996607
- [Derived] Ghosh S, Feagan BG, Ott E, Gasink C, Godwin B, Marano C, Miao Y, Ma T, Loftus EV Jr, Sandborn WJ, Danese S, Abreu MT, Sands BE. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis Through 5 Years in Crohn's Disease and 4 Years in Ulcerative Colitis. J Crohns Colitis. 2024 Aug 6;18(7):1091-1101. doi: 10.1093/ecco-jcc/jjae013. PMID 38310565
- [Derived] Colombel JF, Sands BE, Gasink C, Yeager B, Adedokun OJ, Izanec J, Ma T, Gao LL, Lee SD, Targan SR, Ghosh S, Hanauer SB, Sandborn WJ. Evolution of Symptoms After Ustekinumab Induction Therapy in Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2024 Jan;22(1):144-153.e2. doi: 10.1016/j.cgh.2023.06.014. Epub 2023 Jun 28. PMID 37391056
- [Derived] Dubinsky M, Ma C, Griffith J, Crowell M, Neimark E, Kligys K, O'Connell T. Matching-Adjusted Indirect Comparison Between Risankizumab and Ustekinumab for Induction and Maintenance Treatment of Moderately to Severely Active Crohn's Disease. Adv Ther. 2023 Sep;40(9):3896-3911. doi: 10.1007/s12325-023-02546-6. Epub 2023 Jun 27. PMID 37368103
- [Derived] Adedokun OJ, Xu Z, Gasink C, Kowalski K, Sandborn WJ, Feagan B. Population Pharmacokinetics and Exposure-Response Analyses of Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease. Clin Ther. 2022 Oct;44(10):1336-1355. doi: 10.1016/j.clinthera.2022.08.010. Epub 2022 Sep 21. PMID 36150926
- [Derived] Narula N, Wong ECL, Dulai PS, Marshall JK, Jairath V, Reinisch W. Comparative Effectiveness of Biologics for Endoscopic Healing of the Ileum and Colon in Crohn's Disease. Am J Gastroenterol. 2022 Jul 1;117(7):1106-1117. doi: 10.14309/ajg.0000000000001795. Epub 2022 Apr 15. PMID 35435862
- [Derived] Narula N, Aruljothy A, Wong ECL, Homenauth R, Alshahrani AA, Marshall JK, Reinisch W. The impact of ustekinumab on extraintestinal manifestations of Crohn's disease: A post hoc analysis of the UNITI studies. United European Gastroenterol J. 2021 Jun;9(5):581-589. doi: 10.1002/ueg2.12094. Epub 2021 Jun 2. PMID 34077627
- [Derived] Sandborn WJ, Feagan BG, Danese S, O'Brien CD, Ott E, Marano C, Baker T, Zhou Y, Volger S, Tikhonov I, Gasink C, Sands BE, Ghosh S. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis of Results from Phase 2/3 Studies. Inflamm Bowel Dis. 2021 Jun 15;27(7):994-1007. doi: 10.1093/ibd/izaa236. PMID 32964215
- [Derived] Li K, Friedman JR, Chan D, Pollack P, Yang F, Jacobstein D, Brodmerkel C, Gasink C, Feagan BG, Sandborn WJ, Rutgeerts P, De Hertogh G. Effects of Ustekinumab on Histologic Disease Activity in Patients With Crohn's Disease. Gastroenterology. 2019 Oct;157(4):1019-1031.e7. doi: 10.1053/j.gastro.2019.06.037. Epub 2019 Jul 4. PMID 31279870
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Rutgeerts P, Gasink C, Chan D, Lang Y, Pollack P, Colombel JF, Wolf DC, Jacobstein D, Johanns J, Szapary P, Adedokun OJ, Feagan BG, Sandborn WJ. Efficacy of Ustekinumab for Inducing Endoscopic Healing in Patients With Crohn's Disease. Gastroenterology. 2018 Oct;155(4):1045-1058. doi: 10.1053/j.gastro.2018.06.035. Epub 2018 Aug 29. PMID 29909019
- [Derived] Adedokun OJ, Xu Z, Gasink C, Jacobstein D, Szapary P, Johanns J, Gao LL, Davis HM, Hanauer SB, Feagan BG, Ghosh S, Sandborn WJ. Pharmacokinetics and Exposure Response Relationships of Ustekinumab in Patients With Crohn's Disease. Gastroenterology. 2018 May;154(6):1660-1671. doi: 10.1053/j.gastro.2018.01.043. Epub 2018 Feb 1. PMID 29409871
- [Derived] Hibi T, Imai Y, Murata Y, Matsushima N, Zheng R, Gasink C. Efficacy and safety of ustekinumab in Japanese patients with moderately to severely active Crohn's disease: a subpopulation analysis of phase 3 induction and maintenance studies. Intest Res. 2017 Oct;15(4):475-486. doi: 10.5217/ir.2017.15.4.475. Epub 2017 Oct 23. PMID 29142515
- [Derived] Feagan BG, Sandborn WJ, Gasink C, Jacobstein D, Lang Y, Friedman JR, Blank MA, Johanns J, Gao LL, Miao Y, Adedokun OJ, Sands BE, Hanauer SB, Vermeire S, Targan S, Ghosh S, de Villiers WJ, Colombel JF, Tulassay Z, Seidler U, Salzberg BA, Desreumaux P, Lee SD, Loftus EV Jr, Dieleman LA, Katz S, Rutgeerts P; UNITI-IM-UNITI Study Group. Ustekinumab as Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2016 Nov 17;375(20):1946-1960. doi: 10.1056/NEJMoa1602773. PMID 27959607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 769 participants were randomly assigned to receive study agent. The analyses (efficacy) was based on the 741 participants who were randomized after the study was restarted.
Pre-assignment Details: In November 2011, due to stability issue with the batch of the intravenous (IV) drug (130 mg Ustekinumab) sponsor temporarily suspended dosing of participants with ustekinumab. Later study was restarted with 90 milligram per milliliter (mg/ml).
Groups:
- Placebo: Participants randomized to receive a single dose of Placebo Intravenous (IV) infusion at week 0.
- Ustekinumab 130 Milligram (mg): Participants randomized to receive a single dose of ustekinumab 130 milligram (mg) IV at week 0.
- Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg): Participants randomized to receive tiered ustekinumab dose approximately (~) 6 mg/kg IV at week 0. Ustekinumab 260 mg for participants body weight less than or equal to (< =) 55 kg, ustekinumab 390 mg for weight greater than (>) 55 kg and < = 85 kg and ustekinumab 520 mg for weight > 85 kg.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Started | 256 | 254 | 259
Completed | 244 | 243 | 245
Not Completed | 12 | 11 | 14
Not completed — Withdrawal by Subject | 8 | 6 | 10
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Other | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg) | Total
Number analyzed (Participants) | 256 | 254 | 259 | 769
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.86) | 37.4 (11.74) | 37.2 (12.57) | 37.4 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 153 | 152 | 440
  Male | 121 | 101 | 107 | 329
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 7 | 8 | 21
  Austria | 0 | 0 | 6 | 6
  Belgium | 8 | 12 | 8 | 28
  Brazil | 2 | 0 | 1 | 3
  Canada | 10 | 21 | 21 | 52
  Czech Republic | 2 | 2 | 1 | 5
  Germany | 22 | 14 | 14 | 50
  Denmark | 1 | 3 | 2 | 6
  Spain | 0 | 0 | 2 | 2
  France | 17 | 21 | 29 | 67
  United Kingdom | 21 | 21 | 16 | 58
  Hungary | 1 | 1 | 2 | 4
  Ireland | 0 | 0 | 1 | 1
  Israel | 1 | 2 | 3 | 6
  Italy | 4 | 7 | 8 | 19
  Japan | 18 | 19 | 19 | 56
  South Korea | 1 | 0 | 2 | 3
  Netherlands | 9 | 9 | 14 | 32
  New Zealand | 1 | 1 | 0 | 2
  Poland | 4 | 3 | 4 | 11
  Serbia | 1 | 2 | 1 | 4
  United States | 126 | 108 | 97 | 331
  South Africa | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Week 6
Description: Clinical response at Week 6 was defined as a reduction from baseline in the Crohn's Disease Activity Index score of greater than or equal (>=) 100 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). Participants with a baseline CDAI score of > = 220 to less than or equal (< =) 248 were considered to be in clinical response if a CDAI score of less than (<) 150 was attained. A CDAI score of less than 150 indicates clinical remission. A decrease in CDAI score over time indicates improvement in disease activity.
Time Frame: Baseline and Week 6
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 247 | 245 | 249
participants | 53 | 84 | 84
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 Milligram (mg); Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; 2-sided Cochran-Mantel-Haenszel chi-square test stratified by study region, CDAI score, and initial response to TNF antagonist therapy
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants in Clinical Remission at Week 8
Description: Clinical remission is defined as a CDAI score of less than (<) 150 points at Week 8.
Time Frame: Baseline and Week 8
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 247 | 245 | 249
participants | 18 | 39 | 52
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 Milligram (mg); Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants in Clinical Response at Week 8
Description: Clinical response at Week 8 was defined as a reduction from baseline in the Crohn's Disease Activity Index (CDAI) score of greater than or equal (>=) 100 points. Participants with a baseline CDAI score of > = 220 to less than or equal (< =) 248 were considered to be in clinical response if a CDAI score of less than (<) 150 was attained. A CDAI score of less than 150 indicates clinical remission. A decrease in CDAI score over time indicates improvement in disease activity.
Time Frame: Baseline and Week 8
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 247 | 245 | 249
participants | 50 | 82 | 94
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 Milligram (mg); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Crohn's Disease Activity Index (CDAI) 70-point Response at Week 6
Description: 70-point response is defined as at least 70 points reduction in CDAI score. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline and Week 6
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 247 | 245 | 249
participants | 75 | 113 | 109
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 Milligram (mg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With CDAI 70-point Response at Week 3
Description: as for outcome 4
Time Frame: Baseline and Week 3
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 247 | 245 | 249
participants | 67 | 94 | 101
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 Milligram (mg); Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Week 8 for all participants (for participants who do not enter the maintenance study, adverse events will be collected up to 20 weeks after the study agent administration)
Description: One Participant who was randomized to the placebo group never received study agent and another participant who was randomized to the placebo group actually received ustekinumab and was analyzed in the 130 milligram (mg) ustekinumab group for safety.
Groups:
- Placebo: Participants received a single dose of Placebo Intravenous (IV) infusion at week 0.
- Ustekinumab 130 Milligram (mg): Participants received a single dose of ustekinumab 130 milligram (mg) IV at week 0.
- Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg): Participants received tiered ustekinumab dose approximately (~) 6 mg/kg IV at week 0. Ustekinumab 260 mg for participants body weight less than or equal to (< =) 55 kg, ustekinumab 390 mg for weight greater than (>) 55 kg and < = 85 kg and ustekinumab 520 mg for weight > 85 kg.
Arm/Group | Placebo | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Serious Adverse Events (participants affected / at risk) | 18/254 | 14/255 | 18/259
Other Adverse Events (participants affected / at risk) | 90/254 | 95/255 | 78/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=254) | Ustekinumab 130 Milligram (mg) (N=255) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg) (N=259)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Intracardiac Thrombus (Cardiac disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Colonic Fistula (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 10 | 7 | 5
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Abscess Intestinal (Infections and infestations) | 0 | 1 | 1
Anal Abscess (Infections and infestations) | 1 | 0 | 0
Clostridial Infection (Infections and infestations) | 0 | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0
Infected Fistula (Infections and infestations) | 1 | 0 | 0
Intervertebral Discitis (Infections and infestations) | 0 | 0 | 1
Meningitis Listeria (Infections and infestations) | 0 | 0 | 1
Pelvic Abscess (Infections and infestations) | 0 | 1 | 0
Perineal Abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia Viral (Infections and infestations) | 1 | 0 | 0
Postoperative Abscess (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Vulval Abscess (Infections and infestations) | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Electrolytes Abnormal (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 0 | 0 | 1
Phlebitis Superficial (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=254) | Ustekinumab 130 Milligram (mg) (N=255) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg) (N=259)
Abdominal Pain (Gastrointestinal disorders) | 14 | 10 | 14
Crohn's Disease (Gastrointestinal disorders) | 21 | 8 | 1
Nausea (Gastrointestinal disorders) | 18 | 20 | 15
Fatigue (General disorders) | 13 | 6 | 10
Pyrexia (General disorders) | 14 | 15 | 15
Nasopharyngitis (Infections and infestations) | 14 | 12 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 28 | 15
Headache (Nervous system disorders) | 22 | 20 | 20

LIMITATIONS AND CAVEATS:
The global study was interrupted due to issues with the clinical supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.